CLINICAL TRIAL: NCT05278585
Title: Pacing the Atrium to Confirm or Exclude Pacemaker Indication in TAVI: the PACE-TAVI Registry
Brief Title: Pacing the Atrium to Confirm or Exclude Pacemaker Indication in TAVI
Acronym: PACE-TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Ian Buysschaert, MD PhD, Principal Investigator, AZ Sint-Jan AV
Other Study IDs: version 1 21/02/2022
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RAP TAVI group: All patients in sinus rhythm with TAVI
  Interventions: Procedure: RAP TAVI

INTERVENTIONS:
Procedure: RAP TAVI — All patients undergoing TAVI with no pre-existing pacemaker and in sinus rhythm at the time of the procedure will receive RAP by placing the temporary wire in the right atrium

SUMMARY:
The current observational registry aims to evaluate in patients undergoing TAVI implantation:

1. the positive and negative predictive value for PPM post TAVI of Wenckebach phenomenona (WB) during RAP during the TAVI procedure,
2. baseline and procedural characteristics of TAVI-implantation associated with new conduction abnormalities and need for PPM implantation,
3. peri-procedural safety, in-hospital and 1-month outcomes after TAVI implantation.

DETAILED DESCRIPTION:
The persistent growth in transcatheter aortic valve implantation (TAVI) calls for optimized early discharge programs to handle the increasing patient load. While access site bleeding and stroke rate have decreased with improved technologies and operators' experience, acquired conduction abnormalities necessitating prolonged rhythm-monitoring and permanent pacemaker (PPM) implantation have remained largely unchanged, and even up to 39.9% for some TAVI platforms. Prompt identification of patients necessitating PPM implantation leads to optimal patient care and use of resources. Conversely, prompt identification of patients with low -to no- risk for PPM post TAVI shortens their hospitalization and facilitates early and safe discharge.

Several baseline characteristics such as age, preexistent right bundle branch block (RBBB) and the use of self-expanding valves are associated with post-TAVI PPM implantation, but more practical and clinically more relevant parameters are needed with high negative and positive predictive values that could support clinical decision-making.

En passant rapid atrial pacing (RAP) immediately following TAVI has recently been reported to be a valuable tool in PPM risk stratification. The absence of Wenckebach phenomena post implantation at RAP up to 120/' has a negative predictive value for PPM of 98.7%.2 First use of RAP in routine practice at AZ Sint Jan Brugge can confirm these first results (unpublished data). This technique improves our clinical assessment and identification of low-risk patients for PPM suitable for safe early discharge, as well as high-risk patients requiring further rhythm monitoring and eventual PPM implantation.

The current observational registry aims to evaluate in patients undergoing TAVI implantation:

1. the positive and negative predictive value for PPM post TAVI of Wenckebach phenomenona (WB) during RAP during the TAVI procedure,
2. baseline and procedural characteristics of TAVI-implantation associated with new conduction abnormalities and need for PPM implantation,
3. peri-procedural safety, in-hospital and 1-month outcomes after TAVI implantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients in sinus rhythm with TAVI

Exclusion Criteria:

* Patients in atrial fibrillation at the time of the implantation
* Patients with pre-existent pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients in sinus rhythm undergoing TAVI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Positive and negative predictive value of RAP for PPM implantation post TAVI | 1 month after TAVI
Permanent pacemaker implantation | 1 month after TAVI
New conduction abnormalities | within 1 week after TAVI

SECONDARY OUTCOMES:
Duration of hospitalization | 1 month after TAVI
Echocardiographic changes | 1 month after TAVI
Stroke | 1 month after TAVI
Major vascular bleeding | 1 month after TAVI
New pericardial effusion | 1 month after TAVI
All-cause mortality | 1 month after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Ian Buysschaert, MD, PhD, Principal Investigator — AZ Sint Jan
Locations (12):
- Belgium (12):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - OLV Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - AZ Sint Jan, Bruges
  - CHU Charleroi-Chimay, Charleroi
  - Grand Hôpital de Charleroi, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - Citadelle Hospital, Liège
  - Clinique Saint-Luc Bouge, Namur
  - AZ Delta, Roeselare